CLINICAL TRIAL: NCT06954220
Title: Baduanjin Exercises on Shoulder Dysfunction Post Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005743
Record Dates: First submitted 2025-04-24; First posted 2025-05-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Thyroiditis, Chronic
MeSH Terms: conditions — Thyroiditis, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective Randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin exercises (Experimental): This group included 40 participants post thyroidectomy; they will receive Baduanjin exercises and conservative shoulder care
  Interventions: Other: Baduanjin exercises
- control group (No Intervention): This group included 40 participants post thyroidectomy; they will receive conservative shoulder care

INTERVENTIONS:
Other: Baduanjin exercises — Baduanjin has 8 movement forms, which are relatively less demanding. Assistive equipment is also not necessary during Baduanjin. These advantages make Baduanjin a suitable form of exercise training for post thyroidectomy patients. The movements involved in Baduanjin require the individual to reach beyond the base of support, change the base of support between bilateral and unilateral stance, and perform movements in a sustained squatting posture. These maneuvers challenge balance and require muscle strength to be executed successfully. In 8 movement forms of Baduanjin all include shoulder joint function exercises, thus making Baduanjin a potentially useful method for improving activity level and arm strength.
  Arms: Baduanjin exercises

SUMMARY:
This study will be carried out at the outpatient clinic of the faculty of physical therapy, Cairo university, El Galaa general hosbital after referral from endocrine surgeon. Participants will perform these exercises in a room supervisor physiotherapist.

All participants will sign a written consent form after receiving full information about the purpose of the study, procedure, possible benefits, privacy, and use of data.

DETAILED DESCRIPTION:
This study will investigate the effects of Baduanjin exercises on shoulder dysfunction post thyroidectomy. To assign patients to different treatment groups, a table of random numbers generated by a computer was used. Patients were allocated randomly into two groups using this method. This study will be carried out at the outpatient clinic of the faculty of physical therapy, Cairo University, El Galaa general hospital and National Cancer Institute in Cairo to be treated in the outpatient clinic after referral from endocrine surgeon. Participants will perform these exercises in a room supervisor physiotherapist.

All participants will sign a written consent form after receiving full information about the purpose of the study, procedure, possible benefits, privacy, and use of data.

ELIGIBILITY:
Inclusion Criteria:

* They have the development of the shoulder dysfunction (Range of motion limitation and shoulder pain) (limitation of 20 ≥ ROM in shoulder flexion, abduction, external or internal rotation) after thyroidectomy.
* Patients who were 6 months to 1 year post unilateral neck dissection
* Aged 30- 50 years (at the time of surgery)

Exclusion Criteria:

* they had severe cardiac disease, uncontrolled hypertension and upper extremity problems started Before treatment of thyroid cancer surgery.
* Patients with neurological disease, rheumatologically disease, communication problems, recurrent infections, and history of head or neck malignancy, history of > 1 neck dissection, history of bilateral neck dissection,
* open wounds or incision presence in the region and patients proceeding with chemotherapy (CT) or radiotherapy (RT) were barred

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and disability index (SPADI) | at baseline and at 12 weeks
  It was used to determine the shoulder pain and disability. It comprises of 13 items: a 5 item subscale to evaluate the pain and an 8 item subscale to evaluate the disability. The total score is determined by averaging the pain and disability subscale scores. The SPADI exhibits great construct validity, associating admirably with other district explicit shoulder questionnaires. The translated version of the SPADI in the Arabic language showed excellent internal consistency, with a Cronbach's α values of 0.98, and test retest reliability.the SPADI score ranges from 0 to 100, with higher scores indicating greater shoulder pain and disability

SECONDARY OUTCOMES:
Shoulder range of motion :( active range of motion (ROM)) using Image J | at baseline and at 12 weeks
  The ImageJ, a photograph-based goniometry tool, can measure the angle using images or videos during these exercises. Measurement method using ImageJ during active ROM exercises.Three-dimensional motion capture systems, such as Vicon, have been widely used with increased accuracy . However, as these technologies can be costly and are unavailable in many clinical settings , the ImageJ open-source software is considered particularly for measuring the ROM of the upper limbs during exercise
Total calcium concentration | at baseline and at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No